CLINICAL TRIAL: NCT00464867
Title: Effect of Probiotic on Immunogenicity of Oral Cholera Vaccine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Kyoto University (Other); Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2004-032
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Cholera
Keywords: Bifidobacterium breve; oral whole cell cholera vaccine; immunogenicity; Supplementation with probiotic improves vibriocidal antibody response in 2-5 year old childern given the killed oral cholera vaccine; Supplementation with probiotics results in improving the ASC responses to CT and LPS of V. cholerae O1
MeSH Terms: conditions — Cholera | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Whole cell killed cholera vaccine & probiotic — The oral cholera vaccine Dukoral will be administered to all study participants in two doses,two weeks between doses.Each dose of the formalin inactivated whole cell vaccine contains one mg of recombinant B subunit of cholera toxin(rCTB).The vaccine will be administered in bicarbonate-tartaric acid buffer to counteract the effect of low pH in the stomach.

SUMMARY:
Cholera is a major health problem of many developing countries and marked increase in the prevalence has been seen on all continents in the last decade (WHO 1998). There is a great need for an appropriate vaccine to protect children the principal suffers in endemic countries, from the live threatening consequences of cholera. The B subunit-whole cell killed vaccine (Dukoral) developed in Sweden and used in field trials all over the world. It is licensed in many counties of the world and recommended by WHO. Protective efficacy to the killed vaccine has been demonstrated in adults in Bangladesh as well as in other countries, but less so in children (Clemens et al. 1986). Thus there is an urgency for developing strategies to improve the immunogenicity of vaccines especially for protection of children in cholera endemic countries of the world. Different options for improved cholera vaccines are being considered including new and improved formulations of killed or live oral candidate vaccines (Qadri et al. 2004, Sack et al. 1997, Levine et al. 1993) as well as the use of micronutrient supplementation during the course of immunization (Albert et al. 2003, Karlsen et al. 2003, Qadri et al. 2004). Another option that appears promising is the use of probiotics as adjunct to oral immunization based on the understanding that these agents could improve the mucosal immune responses, both innate and adaptive and help reducing inflammation (Blum and Schiffrin 2003, Fang et al. 2000). A therapeutic as well as preventive role of probiotics has been suggested from results of different studies using different probiotics that have been tested, usually lactic acid producing bacteria such as lactobacillus, Bifidobacterium and Steptococcus species. The supplemention of probiotics to infants may also have a prophylactic effect against acute diarrheal diseases. In pediatric populations, the effect of probiotic agents appears to be most significant against rotavirus diarrhea, suggesting that an immunological mechanism is responsible for the beneficial effects (Saavedra, 2000). In the present proposal we would like to examine if supplementation with the probiotic Bifidobacterium breve has a beneficial role in enhancing the immunogenicity of Dukoral in children. A two cell study will be conducted in which one group of children will be given B. breve every day for four weeks and another group will be given placebo. Two doses of the oral cholera vaccine will be administered at two week interval following initiation of the probiotic/placebo administration. Pre- and post- vaccination blood sample will be collected and assayed for immune response to the vaccine. The frequency and magnitude of the immune response to the vaccine will be compared among the two groups of children to assess whether the probiotic treatment enhances the immune responses to the vaccine. If probiotic supplemenation has a positive effect on the immune response it may be adopted as adjunct to enhance the efficacy of the cholera vaccine in immunization programmes and perhaps also of other enteric vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Children of either sex aged 2-5 years
* Eligible for screening
* Written informed consent from parents
* Free from any chronic illness
* Free from any recent illness
* Apparently healthy without known underlying illness

Exclusion Criteria:

* Children below -2SD of the NCHS reference median
* Severe parasitic and helminthic load
* Presence of enteric pathogen in stool
* History of diarrhoea in the preceding 2 weeks.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2006-01; Primary Completion 2006-01 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Determine vibriocidal antibody response among Bangladeshi children aged 2-5 years given the whole cell killed cholera vaccine | Two years after the enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Firdausi Qadri, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- ICDDR,B, Dhaka, Bangladesh